CLINICAL TRIAL: NCT04888507
Title: A Single Arm, Open-Label Study to Assess the Safety, Efficacy, and Pharmacodynamic Effects of Pozelimab and Cemdisiran Combination Therapy in Patients With Paroxysmal Nocturnal Hemoglobinuria Who Switch From Eculizumab Therapy
Brief Title: Pozelimab and Cemdisiran Combination Therapy in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria Who Switch From Eculizumab Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-20105; 2020-005006-25 (EudraCT Number)
Record Dates: First submitted 2021-04-23; First posted 2021-05-17 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pozelimab+Cemdisiran (Experimental)
  Interventions: Drug: Pozelimab; Drug: Cemdisiran

INTERVENTIONS:
Drug: Pozelimab — Intravenous (IV) loading dose (once) followed after 30 minutes by sub-cutaneous (SC) administration
  Other Names: REGN3918
Drug: Cemdisiran — SC administration
  Other Names: ALN-CC5

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of pozelimab and cemdisiran combination therapy in participants with PNH who switch from eculizumab therapy

The secondary objectives of the study are:

* To evaluate the effect of the combination treatment on the following parameters of intravascular hemolysis: lactate dehydrogenase (LDH) control, breakthrough hemolysis, and inhibition of CH50
* To evaluate the effect of the combination treatment on the stability of LDH during the transition period from eculizumab monotherapy to combination with pozelimab and cemdisiran
* To evaluate the effect of the combination treatment on red blood cell (RBC) transfusion requirements
* To evaluate the effect of the combination treatment on hemoglobin levels
* To evaluate the effect of the combination treatment on clinical outcome assessments (COAs) measuring fatigue and health related quality of life (HRQoL)
* To assess the concentrations of total pozelimab and eculizumab in serum; and total cemdisiran and C5 protein in plasma
* To assess the immunogenicity of pozelimab and cemdisiran
* To assess safety after dose intensification
* To evaluate the long-term safety and efficacy of the combination treatment in an optional open-label extension period (OLEP)

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of paroxysmal nocturnal hemoglobinuria confirmed by a history of high-sensitivity flow cytometry from prior testing
2. Treated with stable (ie, no change in dose or frequency) eculizumab therapy at the labeled dosing regimen or a higher dose and/or more frequently administered than labeled for at least 12 weeks prior to screening visit

Key Exclusion Criteria:

1. History of bone marrow transplantation or receipt of an organ transplant
2. Body weight <40 kg at screening
3. Current plans for modification of the following background concomitant medications, as applicable, during screening and treatment period: erythropoietin, immunosuppressive drugs, corticosteroids, anti-thrombotic agents, anticoagulants, iron supplements, and folic acid as described in the protocol
4. Any use of complement inhibitor therapy other than eculizumab in the 12 weeks prior to the screening visit or planned use during the study
5. Known hypocellular bone marrow based on a history of reduced age-adjusted bone marrow cellularity and/or bone marrow cellularity ≤25%
6. No documented meningococcal vaccination within 5 years prior to screening visit unless it is documented that vaccination has been administered during the screening period and prior to initiation of study treatment
7. Unable to take antibiotics for meningococcal prophylaxis, if required by local standard of care
8. Any active, ongoing infection or a recent infection requiring ongoing systemic treatment with antibiotics, antivirals, or antifungals within 2 weeks of screening or during the screening period
9. Documented positive polymerase chain reaction (PCR) or equivalent test based on regional recommendations for COVID-19 or suspected SARS-CoV-2 infection as described in the protocol
10. Documented history of active, uncontrolled, ongoing systemic autoimmune diseases
11. Recent, unstable medical conditions, excluding PNH and PNH-related complications, within the past 3 months prior to screening visit as described in the protocol
12. Anticipated need for major surgery during the study

NOTE: Other protocol-defined Inclusion/ Exclusion Criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Study Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 7 participants were screened and 6 were enrolled and received study treatment.
Groups:
- Participants With PNH: Participants received cemdisiran by subcutaneous (SC) injection along with their usual dose of eculizumab by intravenous (IV) infusion. After completion of Open Label Treatment Period (OLTP), for participants who willing to continue to receive study treatment, SC pozelimab and cemdisiran Q4W were administered up to 52 weeks during the Open-Label Extension Period (OLEP)
Period: Open-Label Treatment (OLTP) (32 Weeks)
Arm/Group | Participants With PNH
Started | 6
Completed (Completed = Completed OLTP) | 5
Not Completed | 1
Not completed — Adverse Event | 1
Period: Open-Label Extension (OLEP) (52 Weeks)
Arm/Group | Participants With PNH
Started | 5
Completed (Completed = Completed OLEP) | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received any amount of study drug.
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: OLTP: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Up to Day 225
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: OLTP: Percent Change in Lactate Dehydrogenase (LDH) From Pre-treatment to End-of-treatment Period
Time Frame: Screening (Day 1) through Day 225
Population: The full analysis set (FAS) included all enrolled participants who received any amount of study drug and had at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percent change | -0.95 (13.40)

3. Secondary Outcome: OLTP: Percent Change in LDH From Pre-treatment Through Day 29
Time Frame: Screening (Day 1) through Day 29
Population: The FAS included all enrolled participants who received any amount of study drug and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
percent change | 3.61 (35.99)

4. Secondary Outcome: OLTP: Percentage of Participants Who Were Transfusion-free From Baseline Through Week 32
Time Frame: Baseline through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
percentage of participants | 100 [100.0 to 100.0]

5. Secondary Outcome: OLTP: Percentage of Participants Who Were Transfusion-free From Week 4 Through Week 32
Time Frame: Week 4 through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
percentage of participants | 100 [100.0 to 100.0]

6. Secondary Outcome: OLTP: Rate of Red Blood Cell (RBC) Transfusions From Baseline Through Week 32
Description: The rate of units of transfusion for a participant was calculated based on the duration of treatment exposure of the participant.
Time Frame: Baseline through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: transfusions per person-year
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
transfusions per person-year | 0 [NA to NA] — Not calculable due to insufficient number of events.

7. Secondary Outcome: OLTP: Rate of RBC Transfusions From Week 4 Through Week 32
Description: as for outcome 6
Time Frame: Week 4 through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: transfusions per person-year
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
transfusions per person-year | 0 [NA to NA] — Not calculable due to insufficient number of events.

8. Secondary Outcome: OLTP: Number of RBC Units Transfused From Baseline Through Week 32
Time Frame: Baseline through Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
RBC units | 0 (0.0)

9. Secondary Outcome: OLTP: Number of RBC Units Transfused From Week 4 Through Week 32
Time Frame: Week 4 through Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
RBC units | 0 (0.0)

10. Secondary Outcome: OLTP: Percentage of Participants With Breakthrough Hemolysis From Baseline Through Week 32
Description: Breakthrough hemolysis was defined as having an LDH ≥ 2 x upper limit of normal (ULN) and having signs or symptoms.
Time Frame: Baseline through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
percentage of participants | 0.0 [0.0 to 0.0]

11. Secondary Outcome: OLTP: Percentage of Participants With Breakthrough Hemolysis From Week 4 Through Week 32
Description: Breakthrough hemolysis was defined as having an LDH ≥ 2 x ULN and having signs or symptoms.
Time Frame: Week 4 through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
percentage of participants | 0.0 [0.0 to 0.0]

12. Secondary Outcome: OLTP: Percentage of Participants Who Maintained Adequate Control of Hemolysis From Day 1 Through Week 32
Description: Adequate control was defined as LDH ≤ 1.5 x ULN from Day 1 through Week 32.
Time Frame: Day 1 through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 83.3 [53.5 to 100.0]

13. Secondary Outcome: OLTP: Percentage of Participants Who Maintained Adequate Control of Hemolysis From Week 8 Through Week 32
Description: Adequate control was defined as LDH ≤ 1.5 x ULN from Week 8 through Week 32.
Time Frame: Week 8 through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 83.3 [53.5 to 100.0]

14. Secondary Outcome: OLTP: Number of Participants With Adequate Control of Hemolysis at Each Visit
Description: Adequate control at a visit was defined as having LDH ≤1.5 x ULN at that visit.
Time Frame: Days 1, 8, 15, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225
Population: The FAS included all enrolled participants who received any amount of study drug and had at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
Participants
  Day 1 | 6
  Day 8: number analyzed (Participants) | 5
  Day 8 | 5
  Day 15: number analyzed (Participants) | 5
  Day 15 | 5
  Day 29 | 6
  Day 43: number analyzed (Participants) | 5
  Day 43 | 5
  Day 57: number analyzed (Participants) | 5
  Day 57 | 5
  Day 71: number analyzed (Participants) | 5
  Day 71 | 5
  Day 85: number analyzed (Participants) | 5
  Day 85 | 5
  Day 113: number analyzed (Participants) | 4
  Day 113 | 4
  Day 141: number analyzed (Participants) | 5
  Day 141 | 5
  Day 169: number analyzed (Participants) | 4
  Day 169 | 4
  Day 197: number analyzed (Participants) | 3
  Day 197 | 3
  Day 225: number analyzed (Participants) | 5
  Day 225 | 5

15. Secondary Outcome: OLTP: Number of Participants With Normalization of Their LDH at Each Visit
Description: Normalization was defined as LDH ≤ 1.0 x ULN at that visit.
Time Frame: Days 1, 8, 15, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
Participants
  Day 1 | 6
  Day 8: number analyzed (Participants) | 5
  Day 8 | 5
  Day 15: number analyzed (Participants) | 5
  Day 15 | 5
  Day 29 | 6
  Day 43: number analyzed (Participants) | 5
  Day 43 | 5
  Day 57: number analyzed (Participants) | 5
  Day 57 | 4
  Day 71: number analyzed (Participants) | 5
  Day 71 | 5
  Day 85: number analyzed (Participants) | 5
  Day 85 | 4
  Day 113: number analyzed (Participants) | 4
  Day 113 | 4
  Day 141: number analyzed (Participants) | 5
  Day 141 | 5
  Day 169: number analyzed (Participants) | 4
  Day 169 | 4
  Day 197: number analyzed (Participants) | 3
  Day 197 | 3
  Day 225: number analyzed (Participants) | 5
  Day 225 | 5

16. Secondary Outcome: OLTP: Average LDH From Baseline Through Week 32
Description: The trapezoidal rule was used to calculate area under the curve (AUC). Individual mean LDH is defined as AUC divided by (last assessment date of LDH - first assessment date of LDH) of specific period.
Time Frame: Baseline through Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
Units per Liter (U/L) | 227.34 (45.08)

17. Secondary Outcome: OLTP: Average LDH From Week 8 Through Week 32
Description: The trapezoidal rule was used to calculate AUC. Individual mean LDH is defined as AUC divided by (last assessment date of LDH - first assessment date of LDH) of specific period.
Time Frame: Week 8 through Week 32
Population: The FAS included all enrolled participants who received any amount of study drug and had at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
U/L | 223.49 (49.01)

18. Secondary Outcome: OLTP: Percentage of Participants With Hemoglobin Stabilization From Baseline Through Week 32
Description: Hemoglobin stabilization was defined as not receiving an RBC transfusion and having no decrease in hemoglobin level of ≥ 2 grams per deciliter (g/dL).
Time Frame: Baseline through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
percentage of participants | 100 [100.0 to 100.0]

19. Secondary Outcome: OLTP: Percentage of Participants With Hemoglobin Stabilization From Week 4 Through Week 32
Description: Hemoglobin stabilization was defined as not receiving an RBC transfusion and having no decrease in hemoglobin level of ≥ 2 g/dL.
Time Frame: Week 4 through Week 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
percentage of participants | 100 [100.0 to 100.0]

20. Secondary Outcome: OLTP: Change From Baseline in Hemoglobin Levels
Time Frame: Baseline, Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
g/dL | 0.54 (0.60)

21. Secondary Outcome: OLTP: Change From Baseline in Fatigue as Measured by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score
Description: The FACIT-Fatigue is a 13-item, self-reported measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related quality of life (QoL) in participants with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a Likert scale ranging from 0 (not at all) to 4 (very much). Total scores range from 0 to 52, with higher scores indicating a higher quality of life.
Time Frame: Baseline, Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With PNH
Number analyzed (Participants) | 1
score on a scale | -1.0

22. Secondary Outcome: OLTP: Change From Baseline in Health Related Quality of Life (HRQoL) as Measured by the Global Health Status Subscale of the European Organization for Research and Treatment of Cancer (EORTC)- Quality of Life Cancer Patients Questionnaire (QLQ) - 30 Scale
Description: EORTC-QLQ-C30 is a 30-item self-reported questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. The GHS subscale scores ranged from 0 to 100 with higher scores indicating better quality of life.
Time Frame: Baseline, Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With PNH
Number analyzed (Participants) | 1
score on a scale | -8.333

23. Secondary Outcome: OLTP: Change From Baseline in Physical Function (PF) Scores on the EORTC QLQ-C30
Description: EORTC-QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a PF scale. PF subscale scores ranged from 0 to 100 with higher scores indicating better quality of life.
Time Frame: Baseline, Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With PNH
Number analyzed (Participants) | 1
score on a scale | 6.667

24. Secondary Outcome: OLTP: Change From Baseline in Total Complement Hemolytic Activity Assay (CH50)
Description: This assay assessed the activity of the classical pathway of complement to measure C5 activity.
Time Frame: Baseline through Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: International units per mL (IU/mL)
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
International units per mL (IU/mL) | 0.0 (0.0)

25. Secondary Outcome: OLTP and OLEP: Concentration of Total Pozelimab in Serum
Time Frame: Pre-dose Days 28, 56, 84, 112, 140, 168, 196, 224, 392, 588; Post-dose Day 28
Population: The pharmacokinetic (PK) analysis population included all participants who received any amount of study drug and who had at least 1 non-missing result following the first dose of study drug. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
milligrams per liter (mg/L)
  Pre-dose Day 28 | 0 (0)
  15 Minutes Post-dose Day 28 | 1280 (193)
  Pre-dose Day 56 | 333 (48.1)
  Pre-dose Day 84: number analyzed (Participants) | 5
  Pre-dose Day 84 | 189 (54.8)
  Pre-dose Day 112: number analyzed (Participants) | 4
  Pre-dose Day 112 | 121 (57.2)
  Pre-dose Day 140: number analyzed (Participants) | 4
  Pre-dose Day 140 | 102 (40.7)
  Pre-dose Day 168: number analyzed (Participants) | 5
  Pre-dose Day 168 | 70.1 (37.3)
  Pre-dose Day 196: number analyzed (Participants) | 4
  Pre-dose Day 196 | 86.1 (36.6)
  Pre-dose Day 224: number analyzed (Participants) | 5
  Pre-dose Day 224 | 71.7 (41.4)
  Pre-dose Day 392: number analyzed (Participants) | 5
  Pre-dose Day 392 | 53.1 (25.6)
  Pre-dose Day 588: number analyzed (Participants) | 5
  Pre-dose Day 588 | 51.1 (25.6)

26. Secondary Outcome: OLTP: Concentration of Total Eculizumab in Serum
Time Frame: Pre-dose Days 0, 14, 28, 56, 84, 112, 140, 168, 196, 224
Population: The PK analysis population included all participants who received any amount of study drug and who had at least 1 non-missing result following the first dose of study drug. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
mg/L
  Pre-dose Day 0 | 231 (64.5)
  Pre-dose Day 14 | 225 (63.2)
  Pre-dose Day 28 | 242 (59.0)
  Pre-dose Day 56 | 101 (42.9)
  Pre-dose Day 84: number analyzed (Participants) | 5
  Pre-dose Day 84 | 44.4 (38.7)
  Pre-dose Day 112: number analyzed (Participants) | 4
  Pre-dose Day 112 | 22.5 (29.5)
  Pre-dose Day 140: number analyzed (Participants) | 4
  Pre-dose Day 140 | 12.6 (12.5)
  Pre-dose Day 168: number analyzed (Participants) | 5
  Pre-dose Day 168 | 4.23 (6.46)
  Pre-dose Day 224: number analyzed (Participants) | 5
  Pre-dose Day 224 | 0.540 (1.16)

27. Secondary Outcome: OLTP and OLEP: Concentration of Total Cemdisiran in Plasma
Time Frame: Pre-dose and Post-dose Days 0, 84, 196, 224, 588
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL)
  Pre-dose Day 0 | 0 (0)
  Post-dose Day 0 | 139 (45.5)
  Pre-dose Day 84: number analyzed (Participants) | 5
  Pre-dose Day 84 | 0 (0)
  Post-dose Day 84: number analyzed (Participants) | 5
  Post-dose Day 84 | 178 (111)
  Pre-dose Day 196: number analyzed (Participants) | 4
  Pre-dose Day 196 | 0 (0)
  Post-dose Day 196: number analyzed (Participants) | 4
  Post-dose Day 196 | 196 (100)
  Pre-dose Day 224: number analyzed (Participants) | 5
  Pre-dose Day 224 | 0 (0)
  Post-dose Day 224: number analyzed (Participants) | 5
  Post-dose Day 224 | 158 (75.7)
  Pre-dose Day 588: number analyzed (Participants) | 5
  Pre-dose Day 588 | 0 (0)
  Post-dose Day 588: number analyzed (Participants) | 5
  Post-dose Day 588 | 215 (84.8)

28. Secondary Outcome: OLTP and OLEP: Concentration of Total C5 in Plasma
Time Frame: Pre-dose Days 0, 7, 14, 28, 56, 84, 112, 140, 168, 196, 224, 392, 588
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
mg/L
  Pre-dose Day 0 | 320 (64.2)
  Pre-Dose Day 7 | 191 (46.2)
  Pre-dose Day 14 | 118 (28.0)
  Pre-dose Day 28 | 54.5 (14.2)
  Pre-dose Day 56 | 2.77 (6.78)
  Pre-dose Day 84: number analyzed (Participants) | 5
  Pre-dose Day 84 | 2.90 (6.48)
  Pre-dose Day 112: number analyzed (Participants) | 4
  Pre-dose Day 112 | 3.88 (7.75)
  Pre-dose Day 140: number analyzed (Participants) | 5
  Pre-dose Day 140 | 3.10 (6.93)
  Pre-dose Day 168: number analyzed (Participants) | 5
  Pre-dose Day 168 | 4.79 (7.18)
  Pre-dose Day 196: number analyzed (Participants) | 4
  Pre-dose Day 196 | 2.03 (4.05)
  Pre-dose Day 224: number analyzed (Participants) | 5
  Pre-dose Day 224 | 4.96 (7.44)
  Pre-dose Day 392: number analyzed (Participants) | 5
  Pre-dose Day 392 | 5.02 (7.13)
  Pre-dose Day 588: number analyzed (Participants) | 5
  Pre-dose Day 588 | 5.28 (7.44)

29. Secondary Outcome: OLTP: Number of Participants With Pozelimab Anti-drug Antibodies (ADA)
Time Frame: Baseline through Week 32
Population: The ADA analysis set included all participants who received study drug and had at least 1 non-missing ADA result following the first study dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
Participants | 0

30. Secondary Outcome: OLTP: Number of Participants With Cemdisiran ADA
Time Frame: Baseline through Week 32
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 6
Participants | 0

31. Secondary Outcome: OLTP: Number of Participants Who Received Dose Intensification With TEAEs
Time Frame: Baseline through Week 32
Population: No participants required treatment intensification during the study.
Arm/Group | Participants With PNH
Number analyzed (Participants) | 0

32. Secondary Outcome: OLEP: Number of Participants With TEAEs
Time Frame: Day 1 through Week 52 of the OLEP
Population: The OLEP safety analysis set included all participants who participated in the OLEP who received any amount of study drug in the OLEP.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
Participants | 5

33. Secondary Outcome: OLEP: Percent Change in LDH From Day 1 Through Week 24 of the OLEP
Time Frame: Day 1 through Week 24 of the OLEP
Population: The OLEP FAS included all participants who participated in the OLEP who received any amount of study drug in the OLEP and had at least 1 post-baseline assessment in the OLEP.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percent change | -6.17 (9.15)

34. Secondary Outcome: OLEP: Percent Change in LDH From Day 1 Through Week 52 of the OLEP
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percent change | -3.46 (10.94)

35. Secondary Outcome: OLEP: Percentage of Participants Who Were Transfusion-free From Day 1 Through Week 24 of the OLEP
Time Frame: Day 1 through Week 24 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 100 [100.0 to 100.0]

36. Secondary Outcome: OLEP: Percentage of Participants Who Were Transfusion-free From Day 1 Through Week 52 of the OLEP
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 80.0 [44.9 to 100.0]

37. Secondary Outcome: OLEP: Rate of RBC Transfusions From Day 1 Through Week 24 of the OLEP
Description: The rate of units of transfusion for a participants was calculated based on the duration of treatment exposure of the participant.
Time Frame: Day 1 through Week 24 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: transfusions per person-year
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
transfusions per person-year | 0 [NA to NA] — Not calculable due to insufficient number of events.

38. Secondary Outcome: OLEP: Rate of RBC Transfusions From Day 1 Through Week 52 of the OLEP
Description: as for outcome 37
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: transfusions per person-year
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
transfusions per person-year | 0.200 [0.028 to 1.421]

39. Secondary Outcome: OLEP: Number of RBC Units Transfused From Day 1 Through Week 24 of the OLEP
Time Frame: Day 1 through Week 24 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
RBC units | 0 (0.0)

40. Secondary Outcome: OLEP: Number of RBC Units Transfused From Day 1 Through Week 52 of the OLEP
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
RBC units | 0.4 (0.9)

41. Secondary Outcome: OLEP: Percentage of Participants With Breakthrough Hemolysis From Day 1 Through Week 24 of the OLEP
Description: Breakthrough hemolysis was defined as having an LDH ≥ 2 x ULN and having signs or symptoms.
Time Frame: Day 1 through Week 24 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 0.0 [0.0 to 0.0]

42. Secondary Outcome: OLEP: Percentage of Participants With Breakthrough Hemolysis From Day 1 Through Week 52 of the OLEP
Description: Breakthrough hemolysis was defined as having an LDH ≥ 2 x ULN and having signs or symptoms.
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 0.0 [0.0 to 0.0]

43. Secondary Outcome: OLEP: Percentage of Participants Who Maintained Adequate Control of Hemolysis From Day 1 Through Week 24 of the OLEP
Description: Adequate control was defined as LDH ≤ 1.5 x ULN.
Time Frame: Day 1 through Week 24 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 100 [100.0 to 100.0]

44. Secondary Outcome: OLEP: Percentage of Participants Who Maintained Adequate Control of Hemolysis From Day 1 Through Week 52 of the OLEP
Description: Adequate control was defined as LDH ≤ 1.5 x ULN.
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 100 [100.0 to 100.0]

45. Secondary Outcome: OLEP: Number of Participants Who Maintained Adequate Control of Hemolysis at Each Visit in OLEP
Description: Adequate control was defined as LDH ≤ 1.5 x ULN at that visit.
Time Frame: Baseline, Days 57, 113, 169, 225, 281, 365 of the OLEP
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
Participants
  Baseline OLEP | 5
  Day 57 OLEP | 5
  Day 113 OLEP | 5
  Day 169 OLEP | 5
  Day 225 OLEP | 5
  Day 281 OLEP | 5
  Day 365 OLEP | 5

46. Secondary Outcome: OLEP: Number of Participants With Normalization of Their LDH at Each Visit in OLEP
Description: Normalization was defined as LDH ≤ 1.0 x ULN at that visit.
Time Frame: Baseline, Days 57, 113, 169, 225, 281, 365 of the OLEP
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
Participants
  Baseline OLEP | 5
  Day 57 OLEP | 5
  Day 113 OLEP | 5
  Day 169 OLEP | 5
  Day 225 OLEP | 5
  Day 281 OLEP | 5
  Day 365 OLEP | 4

47. Secondary Outcome: OLEP: Average LDH From Day 1 Through Week 24 of the OLEP
Description: as for outcome 17
Time Frame: Day 1 through Week 24 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
U/L | 210.55 (42.64)

48. Secondary Outcome: OLEP: Average LDH From Day 1 Through Week 52 of the OLEP
Description: as for outcome 17
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
U/L | 210.13 (44.91)

49. Secondary Outcome: OLEP: Percentage of Participants With Hemoglobin Stabilization From Day 1 Through Week 24 of the OLEP
Description: as for outcome 19
Time Frame: Day 1 through Week 24 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 100 [100.0 to 100.0]

50. Secondary Outcome: OLEP: Percentage of Participants With Hemoglobin Stabilization From Day 1 Through Week 52 of the OLEP
Description: as for outcome 19
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
percentage of participants | 80.0 [44.9 to 100.0]

51. Secondary Outcome: OLEP: Change From Baseline in Hemoglobin Levels
Time Frame: Day 1 and Week 24 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
g/dL | -0.10 (0.52)

52. Secondary Outcome: OLEP: Change From Baseline in Hemoglobin Levels
Time Frame: Day 1 and Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
g/dL | 0.16 (0.70)

53. Secondary Outcome: OLEP: Change From Baseline in FACIT-Fatigue Score
Description: The FACIT-Fatigue is a 13-item, self-reported measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related quality of life (QoL) in patients with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a Likert scale ranging from 0 (not at all) to 4 (very much). Total scores range from 0 to 52, with higher scores indicating a higher quality of life.
Time Frame: Day 1 and Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
score on a scale | -2.4 (8.7)

54. Secondary Outcome: OLEP: Change From Baseline in HRQoL as Measured by the Global Health Status Subscale of the EORTC-QLQ-30 Scale
Description: EORTC-QLQ-C30 is a 30-item self-reported questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. GHS subscale scores ranged from 0 to 100 with higher scores indicating better quality of life.
Time Frame: Day 1 and Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
score on a scale | -10.000 (18.066)

55. Secondary Outcome: OLEP: Change From Baseline in PF Scores on the EORTC QLQ-C30
Description: as for outcome 23
Time Frame: Day 1 and Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
score on a scale | 0.000 (4.714)

56. Secondary Outcome: OLEP: Change From Baseline in CH50
Description: This assay assessed the activity of the classical pathway of complement to measure C5 activity.
Time Frame: Baseline, Week 16, Week 32, Week 52 of the OLEP
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
IU/mL
  Change at Week 16 | 0.0 (0.0)
  Change at Week 32 | 0.6 (1.3)
  Change at Week 52 | 1.2 (1.8)

57. Secondary Outcome: OLEP: Number of Participants With Pozelimab ADA
Time Frame: Day 1 through Week 52 of the OLEP
Population: The ADA-OLEP analysis set included all participants who received study drug in the OLEP and had at least 1 non-missing ADA result following the first OLEP dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
Participants | 0

58. Secondary Outcome: OLEP: Number of Participants With Cemdisiran ADA
Time Frame: Day 1 through Week 52 of the OLEP
Population: as for outcome 57
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With PNH
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: From signing informed consent up to 84 weeks
Groups:
- OLTP: Participants With PNH; OLEP: Participants With PNH: Participants received cemdisiran by subcutaneous (SC) injection along with their usual dose of eculizumab by intravenous (IV) infusion. After completion of Open Label Treatment Period (OLTP), for participants who willing to continue to receive study treatment, SC pozelimab and cemdisiran Q4W were administered up to 52 weeks during the Open-Label Extension Period (OLEP)
Arm/Group | OLTP: Participants With PNH | OLEP: Participants With PNH
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLTP: Participants With PNH (N=6) | OLEP: Participants With PNH (N=5)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLTP: Participants With PNH (N=6) | OLEP: Participants With PNH (N=5)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 5 (22) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04888507/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT04888507/SAP_001.pdf